CLINICAL TRIAL: NCT02685553
Title: Use of Near Infrared Technology as a Guide in Laparoscopic Resection of Pancreatic Lesions: the COLPAN "Colour-and-resect" Project
Brief Title: Near Infrared Technology and Laparoscopic Resection of Pancreatic Lesions: the COLPAN Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, MD, PhD student, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COLPAN
Record Dates: First submitted 2016-02-14; First posted 2016-02-18 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Neuroendocrine Tumors; Clear Cell Renal Carcinoma; Solid Pseudopapillary Tumors of the Pancreas
MeSH Terms: conditions — Carcinoma, Renal Cell

ARMS (1):
- 1 (Experimental): Use of NIR
  Interventions: Device: NIR

INTERVENTIONS:
Device: NIR — Laparoscopic use of NIR

SUMMARY:
The purpose of this study is to determine whether the use of Near-Infrared Technology can guide the laparoscopic resection of hypervascular neoplasms of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80
* diagnosis of hypervascular pancreatic neoplasms to be treated with laparoscopic surgery

Exclusion Criteria:

* allergy to indocyanine green or other vital stains, indium, shellfish
* chronic kidney insufficiency
* chronic hepatopathy
* hyperthyroidism, thyroid adenomas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of hypervascular pancreatic neoplasms detected intraoperatively by NIR | within the time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona Hospital, Verona, Verona, Italy

REFERENCES:
- [Background] Frangioni JV. In vivo near-infrared fluorescence imaging. Curr Opin Chem Biol. 2003 Oct;7(5):626-34. doi: 10.1016/j.cbpa.2003.08.007. PMID 14580568
- [Background] Verbeek FP, van der Vorst JR, Schaafsma BE, Hutteman M, Bonsing BA, van Leeuwen FW, Frangioni JV, van de Velde CJ, Swijnenburg RJ, Vahrmeijer AL. Image-guided hepatopancreatobiliary surgery using near-infrared fluorescent light. J Hepatobiliary Pancreat Sci. 2012 Nov;19(6):626-37. doi: 10.1007/s00534-012-0534-6. PMID 22790312
- [Background] van der Vorst JR, Vahrmeijer AL, Hutteman M, Bosse T, Smit VT, van de Velde CJ, Frangioni JV, Bonsing BA. Near-infrared fluorescence imaging of a solitary fibrous tumor of the pancreas using methylene blue. World J Gastrointest Surg. 2012 Jul 27;4(7):180-4. doi: 10.4240/wjgs.v4.i7.180. PMID 22905287
- [Background] Winer JH, Choi HS, Gibbs-Strauss SL, Ashitate Y, Colson YL, Frangioni JV. Intraoperative localization of insulinoma and normal pancreas using invisible near-infrared fluorescent light. Ann Surg Oncol. 2010 Apr;17(4):1094-100. doi: 10.1245/s10434-009-0868-8. Epub 2009 Dec 22. PMID 20033320